CLINICAL TRIAL: NCT06661044
Title: Exploiting Human Microbiota-associated in Vivo Models for Mechanistic Studies to Understand the Benefits of Dietary Fibre Supplementation in Patients With Prostate Cancer
Brief Title: Understanding the Benefits of Dietary Fibre Supplementation in Patients With Prostate Cancer
Acronym: EVENTIDE
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-054-24; 556 (Other Grant/Funding Number: NHS Grampian Charity, UK)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: Prostate cancer; Dietary fibre; Faecal microbiota transplant; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples will be stored until the study has been completed and then for further 5 years to allow for potential additional analysis in future ethically reviewed and approved studies. Anonymised 16S rRNA gene-based gut microbiota profiling sequence data will be uploaded to a publicly accessible data repository prior to publication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The digestive tract (large intestine) contains microorganisms that digest complex carbohydrates in food to produce chemical substances which are beneficial to human health. The population of these microorganisms in faeces (stool samples) could be used to diagnose the health status of a person and this can be changed with the use of antibiotics, diet, radiotherapy or infection.

Dietary fibre supplements can help provide nutrients for the beneficial bacteria from the large intestine to produce useful chemicals that may delay growth or even shrink prostate cancer in patients.

The investigators will feed mice diets containing several dietary fibres (including inulin, pectin and hemp hull) and also faeces from healthy male human volunteers over 60 years old to see what effect this has on the makeup of the bacteria in their gut and the resulting beneficial metabolites (chemicals). For this work, the research team need to obtain four to six fresh faecal samples on the same day, so that these can be mixed fresh and stored for use as faecal microbiota transplant (FMT) in the mice.

The researchers will then test how altering the gut microorganisms with faeces and dietary fibre supplements can influence the growth of prostate cancer cell tumours in mice. The investigators expect to see an effect of the fibres in promoting beneficial bacteria and in shrinking the tumours.

This work will allow the investigators to identify dietary fibres that could be used in nutritional therapies for management of prostate cancer patients in future.

DETAILED DESCRIPTION:
Prostate cancer is the commonest cancer in men and the fifth most common cause of cancer-related deaths globally. Increased prostate-specific antigen (PSA) screening and longer life expectancies in men have resulted in a substantial increase in the incidence and prevalence of prostate cancer in older men. Between 2021 and 2022, over 50,000 newly diagnosed cases of prostate cancer were reported in the UK, representing a 27% increase in incidence compared to 2019 and causing over 16,000 deaths.

Prostate cancer in its initial stages maybe asymptomatic and progresses slowly, meaning that some men do not need immediate active treatment but can be monitored on 'active surveillance'. Active surveillance was developed as an approach to addressing overtreatment; by delaying or preventing unnecessary definitive treatment, typically surgical removal of the prostate (radical prostatectomy, RP) or radical radiotherapy to the prostate (RT), and their related complications. It involves routine monitoring of PSA levels, medical imaging, digital rectal exams, and prostate biopsies and is recommended for prostate cancer patients with a low risk of developing aggressive tumours.

The process of active surveillance can be quite stressful for some patients and many of these patients are eager to do everything they can to slow the progression of their disease, including making lifestyle changes such as changing their diet and doing physical exercise.

Diet influences the diversity of the microbiota (archaea, bacteria, fungi and viruses) in the gastrointestinal tract. The gut microbiota play crucial functions in metabolic and regulatory processes that impact the body's immunity and disease development. One can increase the consumption of dietary fibre by providing supplements in powder or capsule form, where the dose administered can be controlled. When these dietary fibres are eaten, commensal colonic bacteria ferment them to produce metabolites, including short-chain fatty acids (SCFAs) which can have anti-tumour effects.

This study team and other researchers have reported the effect of the soluble dietary fibre inulin in delaying tumour growth in mice compared to low dietary fibre intake, in a range of tumour types (including bladder and colorectal cancers). Pectin has also been reported to have health benefits such as maintaining the intestinal barrier, improving physical bowel function and reducing glucose and cholesterol absorption. Apple pectin has also been shown to induce apoptosis in colorectal cancer cells.

UK fibre intake at a population level is well below the recommended levels of 30 g per day, with only 9% of adults meeting recommended intakes.

According to a US population-based study, higher fibre intake was inversely associated with prostate cancer aggressiveness and in an intervention study with modified citrus pectin, 78% of men with non-metastatic prostate cancer who had biochemically relapsed responded to therapy: 58% showed decreased PSA and 75% showed improvement in PSA doubling time (p=0.003).

Inulin and pectin are purified soluble fibres from chicory root, citrus, apple and other plants; in contrast, hemp hull is a rich source of whole fibre which also contains bioactive chemicals including flavonoids, proanthocyanidins and phenolic acids. It has been previously reported to have biological activities such as immune-modulating, anti-inflammatory and antineoplastic properties in different cancer cells. Furthermore, hemp hull is a rich source of phytic acid which releases myo-inositol in the human intestine by the activity of microbial phytases. Myoinositol supplementation significantly decreased triglycerides; men with elevated triglycerides might be at increased risk of developing prostate cancer or recurrence following surgery. Therefore, the consumption of whole fibres would bring additional benefits in the prevention of prostate cancer. Preliminary animal studies demonstrated that dietary phytic acid increased the production of microbial short-chain fatty acids (SCFA), including propionate and butyrate, with changes in microbial composition.

Hemp hull is a sustainable fibre source, from a carbon-neutral crop promoting agricultural biodiversity which can help meet dietary fibre intake recommendations. Hemp hulls (obtained after seed decortication) contain 74% fibre which can be milled into hemp hull flour.

Another method to improve tumour control by modifying the gut microbiota, which could be combined with dietary fibre supplementation, is via faecal microbiota transplantation (FMT). This method involves transferring faecal bacteria and other microorganisms from a healthy individual into another person to directly alter the recipient's microbial composition and provide a health benefit. There is increasing interest in the use of FMT for gastrointestinal infections and inflammatory diseases, as well as extraintestinal conditions including autoimmune and metabolic disorders such as cancer, diabetes and non-alcoholic fatty liver disease. In another study, FMT was administered with cancer immunotherapy drugs (nivolumab or pembrolizumab) to mice and enhanced the activity of these drugs in controlling the growth of MCA-205 sarcoma tumours. Also, in a phase I trial, 65% of all patients who received a faecal transplant successfully acquired similarity to the donor microbiomes and experienced an enrichment of immunogenic bacteria and a loss of deleterious bacteria following FMT.

ELIGIBILITY:
Inclusion Criteria:

* Men (biologically male) over 60 years old.
* Regularly pass a bowel motion at least daily.
* Able to attend the Rowett Institute for consent procedure and able to arrange delivery of fresh faecal sample to the Rowett Institute on the required study day.

Exclusion Criteria:

* Living with cancer/on active cancer treatment.
* Active ulcerative colitis or Crohn's disease.
* Antibiotic therapy within previous 3 months.
* Diarrhoea from recent foreign travel.
* Known HIV or Hepatitis B positive.
* Working directly on specific study for which samples are required.
* Line managed or supervised by PI of study.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is interested in looking at prostate cancer and accepts only biological male volunteers.
Study Population: The investigators will also invite men over 60 years who are staff at the University of Aberdeen, via All Staff mailing lists (including SMMSN and Rowett) and the University's weekly News Update and small ads.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
16S rRNA gene sequencing | December 2024 to October 2025
  The investigators will extract bacterial DNA for 16S rRNA gene sequencing analysis to compare the baseline microbial community of volunteers to that of the mice microbiota after faecal microbiota transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Kiltie, MA, DN, DSc, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not appropriate

REFERENCES:
- [Result] Routy B, Lenehan JG, Miller WH Jr, Jamal R, Messaoudene M, Daisley BA, Hes C, Al KF, Martinez-Gili L, Puncochar M, Ernst S, Logan D, Belanger K, Esfahani K, Richard C, Ninkov M, Piccinno G, Armanini F, Pinto F, Krishnamoorthy M, Figueredo R, Thebault P, Takis P, Magrill J, Ramsay L, Derosa L, Marchesi JR, Parvathy SN, Elkrief A, Watson IR, Lapointe R, Segata N, Haeryfar SMM, Mullish BH, Silverman MS, Burton JP, Maleki Vareki S. Fecal microbiota transplantation plus anti-PD-1 immunotherapy in advanced melanoma: a phase I trial. Nat Med. 2023 Aug;29(8):2121-2132. doi: 10.1038/s41591-023-02453-x. Epub 2023 Jul 6. PMID 37414899
- [Result] Smits LP, Bouter KE, de Vos WM, Borody TJ, Nieuwdorp M. Therapeutic potential of fecal microbiota transplantation. Gastroenterology. 2013 Nov;145(5):946-53. doi: 10.1053/j.gastro.2013.08.058. Epub 2013 Sep 7. PMID 24018052
- [Result] Bui TPN, Manneras-Holm L, Puschmann R, Wu H, Troise AD, Nijsse B, Boeren S, Backhed F, Fiedler D, deVos WM. Conversion of dietary inositol into propionate and acetate by commensal Anaerostipes associates with host health. Nat Commun. 2021 Aug 10;12(1):4798. doi: 10.1038/s41467-021-25081-w. PMID 34376656
- [Result] Allott EH, Howard LE, Cooperberg MR, Kane CJ, Aronson WJ, Terris MK, Amling CL, Freedland SJ. Serum lipid profile and risk of prostate cancer recurrence: Results from the SEARCH database. Cancer Epidemiol Biomarkers Prev. 2014 Nov;23(11):2349-56. doi: 10.1158/1055-9965.EPI-14-0458. Epub 2014 Oct 10. PMID 25304929
- [Result] Zhu S, Hu X, Fan Y. Association of triglyceride levels and prostate cancer: a Mendelian randomization study. BMC Urol. 2022 Oct 31;22(1):167. doi: 10.1186/s12894-022-01120-6. PMID 36316671
- [Result] Tabrizi R, Ostadmohammadi V, Lankarani KB, Peymani P, Akbari M, Kolahdooz F, Asemi Z. The effects of inositol supplementation on lipid profiles among patients with metabolic diseases: a systematic review and meta-analysis of randomized controlled trials. Lipids Health Dis. 2018 May 24;17(1):123. doi: 10.1186/s12944-018-0779-4. PMID 29793496
- [Result] Ligresti A, Moriello AS, Starowicz K, Matias I, Pisanti S, De Petrocellis L, Laezza C, Portella G, Bifulco M, Di Marzo V. Antitumor activity of plant cannabinoids with emphasis on the effect of cannabidiol on human breast carcinoma. J Pharmacol Exp Ther. 2006 Sep;318(3):1375-87. doi: 10.1124/jpet.106.105247. Epub 2006 May 25. PMID 16728591
- [Result] Keizman D, Frenkel M, Peer A, Kushnir I, Rosenbaum E, Sarid D, Leibovitch I, Mano R, Yossepowitch O, Margel D, Wolf I, Geva R, Dresler H, Rouvinov K, Rapoport N, Eliaz I. Modified Citrus Pectin Treatment in Non-Metastatic Biochemically Relapsed Prostate Cancer: Results of a Prospective Phase II Study. Nutrients. 2021 Nov 28;13(12):4295. doi: 10.3390/nu13124295. PMID 34959847
- [Result] Tabung F, Steck SE, Su LJ, Mohler JL, Fontham ET, Bensen JT, Hebert JR, Zhang H, Arab L. Intake of grains and dietary fiber and prostate cancer aggressiveness by race. Prostate Cancer. 2012;2012:323296. doi: 10.1155/2012/323296. Epub 2012 Nov 13. PMID 23213538
- [Result] Blanco-Perez F, Steigerwald H, Schulke S, Vieths S, Toda M, Scheurer S. The Dietary Fiber Pectin: Health Benefits and Potential for the Treatment of Allergies by Modulation of Gut Microbiota. Curr Allergy Asthma Rep. 2021 Sep 10;21(10):43. doi: 10.1007/s11882-021-01020-z. PMID 34505973
- [Result] Ewaschuk JB, Dieleman LA. Probiotics and prebiotics in chronic inflammatory bowel diseases. World J Gastroenterol. 2006 Oct 7;12(37):5941-50. doi: 10.3748/wjg.v12.i37.5941. PMID 17009391
- [Result] Li Y, Elmen L, Segota I, Xian Y, Tinoco R, Feng Y, Fujita Y, Segura Munoz RR, Schmaltz R, Bradley LM, Ramer-Tait A, Zarecki R, Long T, Peterson SN, Ronai ZA. Prebiotic-Induced Anti-tumor Immunity Attenuates Tumor Growth. Cell Rep. 2020 Feb 11;30(6):1753-1766.e6. doi: 10.1016/j.celrep.2020.01.035. PMID 32049008
- [Result] Then CK, Paillas S, Wang X, Hampson A, Kiltie AE. Association of Bacteroides acidifaciens relative abundance with high-fibre diet-associated radiosensitisation. BMC Biol. 2020 Aug 19;18(1):102. doi: 10.1186/s12915-020-00836-x. PMID 32811478
- [Result] de Vos II, Luiting HB, Roobol MJ. Active Surveillance for Prostate Cancer: Past, Current, and Future Trends. J Pers Med. 2023 Apr 3;13(4):629. doi: 10.3390/jpm13040629. PMID 37109015
- [Result] Siegel DA, O'Neil ME, Richards TB, Dowling NF, Weir HK. Prostate Cancer Incidence and Survival, by Stage and Race/Ethnicity - United States, 2001-2017. MMWR Morb Mortal Wkly Rep. 2020 Oct 16;69(41):1473-1480. doi: 10.15585/mmwr.mm6941a1. PMID 33056955
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- See also: NDNS: results from years 9 to 11 (2016 to 2017 and 2018 to 2019) — https://www.gov.uk/government/statistics/ndns-results-from-years-9-to-11-2016-to-2017-and-2018-to-2019
- See also: National Prostate Cancer Audit (NPCA), NPCA State of the Nation Report — https://www.npca.org.uk/reports/npca-state-of-the-nation-report